CLINICAL TRIAL: NCT00326040
Title: A Study of the Glaukos Trabecular Micro-Bypass Stent in Refractory Open Angle Glaucoma Subjects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Head of Clinical Affairs, Glaukos Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-001A
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle; Glaucoma; Refractory; Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Device: Glaucoma Surgery

INTERVENTIONS:
Device: Glaucoma Surgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the iStent trabecular micro-bypass stent in reducing intraocular pressure (IOP) in refractory open-angle glaucoma subjects.

DETAILED DESCRIPTION:
Glaukos Corporation conducted a clinical research study at multiple (approximately 7) investigational sites within Europe.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subject on maximally tolerated medical therapy or where noncompliance with medication has been document
* Subject has failed a conventional glaucoma surgical procedure. (trabeculectomy, Trabeculoplasty(ALT), viscocanalostomy, collagen implant)

Exclusion Criteria:

* Angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Affairs, Study Director — Glaukos Corporation
Locations (7):
- Germany (2):
  - University of Cologne, Cologne
  - Klinik für Augenheilkunde, Neubradenbrug
- Italy (2):
  - University Eye Clinic, Genova
  - Instituto di Oftalmologia, Parma
- Ophthalmic Clinic, Rotterdam, Netherlands
- Spain (2):
  - Hospital Clínico San Carlos, Madrid
  - Instituo Oftalmologico de Aragon, Zaragoza